CLINICAL TRIAL: NCT00682760
Title: Double-Blind, Randomized, Phase 3, Comparative Study of a New Botulinum Toxin Type A Versus Botox in the Treatment of Essential Blepharospasm
Brief Title: Comparison of Korean Botulinum Toxin Type A Versus Botox in the Treatment of Essential Blepharospasm
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pacific Pharmaceuticals (Industry)
Responsible Party: KI-YOON, KIM/ CRA of Pacific Pharm, Department of ophthalmology, Yonsei university College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Meditoxin_Botox; Meditoxin-05-01
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Blepharospasm
Keywords: Botulinum Toxin Type A; Blepharospasm
MeSH Terms: conditions — Blepharospasm | interventions — 26S proteasome non-ATPase regulatory subunit 13; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Korean botulinum toxin A treatment
  Interventions: Drug: Korean Botulinum toxin type A (KbtxA) and Botox injection
- 2 (Placebo Comparator): Botox treatment
  Interventions: Drug: Korean Botulinum toxin type A (KbtxA) and Botox injection

INTERVENTIONS:
Drug: Korean Botulinum toxin type A (KbtxA) and Botox injection — Each vial of Botox and KbtxA contained 100 U of BTX-A in a sterile vacuum-derived form without preservatives. Each vial of KbtxA was identical to the placebo (Botox) vial, and all vials were reconstituted with 2.0 mL of 0.9% sterile nonpreserved saline solution to a final dilution of 5 U /0.1 mL. The dose of BTX-A per injection site was 2.5 U to 5 U, and the location, number of injection sites. Using a 30-gauge needle, injections were angled away from the center of lid to reduce the risk of spread into the levator muscle. Injection sites include the upper medial and lateral eyelid margins, lower lateral lid margins, and above the eyebrow.
  Other Names: arm1 ; Meditoxin or Neuronox

SUMMARY:
To compare the efficacy and safety of Korean botulinum toxin A (KbtxA, Pacific Pharmaceuticals, Korea) against Botox in the treatment of essential blepharospasm, we performed a double-blinded, randomized, comparative trial comparing KbtxA and Botox for treatment of blepharospasm in 60 patients of the intention to treat population and 52 patients (26 patients from each group) of the per protocol population. The improvement of severity of spasm (SS) at 4 weeks post-injection as a primary efficacy outcome, qualifying non inferiority to the control group, Changes in eyelid closure force (CF) and functional visual status (FVS) after injection for secondary efficacy outcomes, and adverse effects for safety evaluation. Improvement of SS was noted in 90.3% of the KbtxA group and 86.2% of the Botox group. There were no significant differences between treatment groups in the changes of CF and FVS after injection (p>0.05). Adverse effects developed in 16.1% of the KbtxA group and 27.6% of the Botox group, but no serious adverse events were found in either group. KbtxA was not inferior to Botox in treatment efficacy and was clinically safe with no serious adverse effects when used to treat essential blepharospasm.

DETAILED DESCRIPTION:
Severity of spasm was graded clinically from grade 0 to 4. Primary efficacy outcome was assessed as the number (%) of patients with improved SS of more than 1 score at 4 weeks post-injection. Secondary efficacy outcome measures included the change in scores from baseline on the SS, closing force of eyelids, and functional visual status at 4 weeks post-injection. The duration of action (days), the time interval between injection and the moment that the patient felt the need for retreatment were also assessed as secondary efficacy outcomes.

The number (%) of patients with improvement of SS (primary efficacy outcome) and the change in scores from baseline at 4 weeks post-injection on the severity of spasm, closing force of eyelids, and functional visual status scores were not different between the KbtxA and Botox groups in the analysis of both the ITT and PP populations. Also, the duration of action was similar following KbtxA and Botox injections (two sample t-test, p=0.835). For the non-inferiority trial on primary efficacy outcome, KbtxA was not inferior to Botox in either the ITT or PP populations, as the lower limit of the 95% confidence interval (-1.76% for ITT, -1.64% for PP) was over the -15% threshold.

ELIGIBILITY:
Inclusion Criteria:

* All patients, aged between 18 and 75 years old, had confirmed diagnoses of bilateral essential blepharospasm.
* The patients were recruited from two botulinum toxin clinics (Yonsei University and Chung-Ang University, Seoul, Korea) from October 18, 2005 until February 21, 2006.

Exclusion Criteria:

* Patients were not eligible for inclusion in the study if they

  * had undergone either myectomy or neurectomy
  * had received anti-spastic, muscle relaxant medication within 1 month of study entry
  * had been injected previously with BTX-A within 3 months of study entry
  * had any muscle disorder
* Women with positive urine pregnancy test, or who were pregnant or lactating were also excluded from the study.
* In addition, patients who had shown hypersensitivity to BTX-A previously were not eligible for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-10; Primary Completion 2006-02 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The improvement of severity of spasm at 4 weeks post-injection as a primary efficacy outcome, qualifying non inferiority to the control group | at 4 weeks post-injection

SECONDARY OUTCOMES:
Changes in eyelid closure force and functional visual status after injection for secondary efficacy outcomes | at 4 weeks post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Sang Y Lee, MD, phD, Principal Investigator — Yonsei University
Locations (1):
- Sang Yeul Lee, Seoul, South Korea

REFERENCES:
- [Background] Stone AV, Ma J, Whitlock PW, Koman LA, Smith TL, Smith BP, Callahan MF. Effects of Botox and Neuronox on muscle force generation in mice. J Orthop Res. 2007 Dec;25(12):1658-64. doi: 10.1002/jor.20450. PMID 17600825
- [Derived] Yoon JS, Kim JC, Lee SY. Double-blind, randomized, comparative study of Meditoxin versus Botox in the treatment of essential blepharospasm. Korean J Ophthalmol. 2009 Sep;23(3):137-41. doi: 10.3341/kjo.2009.23.3.137. Epub 2009 Sep 8. PMID 19794937